CLINICAL TRIAL: NCT06595095
Title: The Correlation Characteristics Between Mental Health and Gut Microbiota of College Students in Qingyuan Vocational Education City
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yan He, Professor, Zhujiang Hospital
Other Study IDs: zhujiangjy-20240701
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy individuals
- Anxious Individuals
- Depressive Individuals

SUMMARY:
The goal of this observational study is to learn about the mental health status and gut microbiota characteristics of college students in Qingyuan Vocational Education City. The main question it aims to answer is:

How is the mental condition of college students in Qingyuan Vocational Education City? Is there a correlation between the mental condition and the microbial characteristics of college students in Qingyuan Vocational Education City? Participants will answer online survey questions about their demographic characteristics, disease history, gastrointestinal status, lifestyle habits, and psychological health information. 200 participants from each of the following groups will be included: healthy individuals, anxious Individuals and depressive Individuals. Fecal samples will be collected for microbiome testing and analysis to obtain their microbial characteristics and to analyze the impact of mental health status on microbial changes.

ELIGIBILITY:
Inclusion Criteria:

Healthy Individuals:

1. Ages 18 to 25 years old.
2. Resident in the local area for more than one month.
3. No obvious signs or symptoms of disease.
4. Good psychological condition.
5. College students currently enrolled in Qingyuan Vocational Education City.
6. Having signed an informed consent form, willing to provide relevant survey information and fecal samples.

Anxious Individuals:

1. Ages 18 to 25 years old.
2. Resident in the local area for more than one month.
3. Self-rating anxiety scale score greater than or equal to 50.
4. College students currently enrolled in Qingyuan Vocational Education City.
5. Having signed an informed consent form, willing to provide relevant survey information and fecal samples.

Depressive Individuals:

1. Ages 18 to 25 years old.
2. Resident in the local area for more than one month.
3. Self-rating depression scale score greater than or equal to 53.
4. College students currently enrolled in Qingyuan Vocational Education City.
5. Having signed an informed consent form, willing to provide relevant survey information and fecal samples.

Exclusion Criteria:

1.Pregnant and Lactating Women.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: College students aged 18-25 years old at Qingyuan Vocational Education City
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Microbiota Characteristic Data | 2024.10-2025.9
  The characteristics of microbiota include composition, abundance, and diversity, etc.

SECONDARY OUTCOMES:
general information of participants by questionnaire | 2024.10-2025.9
  The general information of participants will be collected through questionnaire, which includes demographic characteristics, disease history, gastrointestinal status, and lifestyle habits.
Self-Rating Anxiety Scale SAS | 2024.10-2025.9
  Participants will fill out this scale. The total score of the scale is 25-100. The cut-off value of SAS standard score is 50 points, with 50-59 points indicating mild anxiety, 60-69 points indicating moderate anxiety, and 69 points or above indicating severe anxiety.
Self-rating depression scale SDS | 2024.10-2025.9
  Participants will fill out this scale. The total score of the scale is 25-100, with 53 points indicating normal, 53-62 points indicating mild depression, 63-72 points indicating moderate depression, and above 72 points indicating severe depression.
Pittsburgh sleep quality index PSQI | 2024.10-2025.9
  Participants will fill out this scale. The total score of the scale is 0-21 points and can be divided into three levels. PSQI score ≤ 4 indicates good sleep quality, PSQI score ≤ 7 indicates average sleep quality, and PSQI score ≥ 8 indicates poor sleep quality (sleep disorders). Higher PSQI total scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Yan He, Doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang hospital of southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No